CLINICAL TRIAL: NCT04557657
Title: Evaluation of Marginal Integrity Using Modified USPHS Criteria of a Bioactive Cement in Comparison to Resin Cement in Cementation of Indirect Composite Blocks: A Randomized Clinical Trial 12 Month Follow up
Brief Title: Evaluation of Marginal Integrity Using Bioactive Cement Incementation of Indirect Composite Blocks
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Sherif, Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEBD-CU-2019-07-17
Record Dates: First submitted 2020-09-11; First posted 2020-09-21 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Resin Cement
Keywords: Composite blocks; Cad/Cam; Cerec
MeSH Terms: interventions — Resin Cements

STUDY DESIGN:
Intervention Model Description: 36 volunteer assigned randomly into 2 equal groups of 18
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group Resin cement (Experimental): Control group Using resin cement
  Interventions: Drug: Resin Cement
- Intervention Group Active Cement (Active Comparator): Intervention Group Using active cement bio activa
  Interventions: Drug: Active bio Activa

INTERVENTIONS:
Drug: Active bio Activa — Cement that release fluoride
  Other Names: Active Cement Pulpodent
  Arms: Intervention Group Active Cement
Drug: Resin Cement — Resin Cement Convinonal
  Arms: Control Group Resin cement

SUMMARY:
The aim of this study is to evaluate of marginal integrity of indirect composite restoration after cementation by a bioactive cement in comparison to dual cure resin cement using Modified USPHS criteria

DETAILED DESCRIPTION:
The study will be conducted in Conservative Dentistry Department, Faculty of Dentistry, Cairo University, The operator in charge will be: Mohamed Sherif . The researcher will bear ultimate responsibility for all activities associated with the conduct of a research project including recruitment of patients, explaining and performing the procedures to them,A total of 36 volunteer patients with Patients with badly broken vital teeth with minimum of two remaining walls. Patients will be randomly divided into two groups according to type of cement (S) where in group S1, Restoration will be cemented with resin cement ; while group S2,Restoration will be cemented with active cement. Each restoration will be assessed after three, six months and one year using modified USPH Criteria Marginal Discoloration, Recurrent Caries and Marginal Chipping with scale of Alpha and non alpha

ELIGIBILITY:
Inclusion Criteria:

* Patients with badly broken vital teeth with minimum of two remaining walls
* Adult Males or female 16- 65 years old
* Good oral hygiene measures with a good gingival condition
* Cooperative patients approving to participate in the study
* Free of any medical condition that interfere with procedures

Exclusion Criteria:

* Patients with a compromised medical history.
* Severe or active periodontal disease
* Endodontically treated teeth
* Severe medical complications Lack of compliance

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Marginal Discoloration | 12 Months
  Check Marginal Discoloration Using Modified USPH criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, EL Manial, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Individual patient Data can be shared Upon request
Supporting Information: Study Protocol
Time Frame: 1 Year
Access Criteria: Mail